CLINICAL TRIAL: NCT02727608
Title: Induction With Complement Inhibitor Eculizumab in Clinical Islet Transplantation
Brief Title: Complement Inhibitor Eculizumab in Clinical Islet Transplantation
Acronym: ICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICC version 2; 2014-005421-12 (EudraCT Number)
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): Intravenous infusion
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Intravenous infusion (1200 mg) over 35 minutes. Consecutive infusions (900 mg) on Days 1, 7 and 14.
  Other Names: Soliris

SUMMARY:
This is a dual centre, single arm, exploratory study of the possibility to use eculizumab (Soliris) to prevent/reduce destruction of islets of Langerhans after portal infusion of the islets in patients with diabetics accepted for islet transplant.

DETAILED DESCRIPTION:
This is a dual centre, single arm, exploratory study of the possibility to use eculizumab (Soliris) to prevent/reduce destruction of islets of Langerhans after portal infusion of the islets in patients with diabetics accepted for islet transplant. Ten patients from 2 centres (Uppsala University Hospital and Karolinska University Hospital in Stockholm) will be transplanted. The purpose of the study is to investigate if selective complement inhibition by eculizumab combined with standard anticoagulation during and after transplantation can further reduce the extent of early tissue loss after portal infusion of islets.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 65 years of age
* Patients able to provide written informed consent
* Absent stimulated c-peptide (< 0.1 nmol/L). This includes also previously islet-transplanted patients with no detectable c-peptide.
* Patients at fear of severe hypoglycemia
* Female patients of child bearing potential must have a negative pregnancy test (s-β-HCG) and must be practicing an effective, reliable medical accepted contraceptive regimen while on eculizumab treatment and to study end at 75 days.
* Patients vaccinated against Neisseria meningitides or patients accepting adequate antibiotic prophylaxis

Exclusion Criteria:

* Body mass index > 30 kg/m2
* Untreated proliferative diabetes retinopathy
* Recipient of any other concomitant organ transplantation - Glomerular filtration rate < 50 mL/min before first islet transplantation
* Positive T-cell cross-matching by Complement Depending Cytotoxicity (CDC)
* Pregnancy or lactating
* Active ongoing infection, bacterial or viral
* Unresolved meningococcal disease
* Known bleeding disorder
* Known complement disorder
* Have received any other investigational drug within 30 days before inclusion
* History of drug or alcohol abuse within the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Increased survival of ICC´s transplanted as measured by peak c-peptide | During and within two hours post infusion (day 0).
  Determined by PET-scan of 2-deoxy-27fluoro-D-glucose (18F) (FDG)-labelled islets infused in the portal vein.

SECONDARY OUTCOMES:
Effect of eculizumab on instant blood mediated inflammatory reaction (IBMIR) as determined by complement activation. | At the end of infusion and 1 and 2 h post start of infusion (day 0).
  Extent of early tissue loss
Monitoring of islet-function and survival. | 14, 30 and 75 days post-transplant.
  Evaluation of insulin-independency, the extent of reduction of baseline insulin requirement, continuous glucose monitoring system (CGMS) performance, HbA1c, number of hypoglycemic events per week.
Adverse events (AEs) and serious adverse events (SAEs) | From start of infusion until 75 days post-transplant.
  Will be assigned Medical Drug Regulatory Activities (MedDRA) preferred terms and tabulated as incidence rate
Patient and graft survival at 75 days post treatment. | From start of infusion until 75 days post-transplant.
  Graft survival is measured by measurable stimulated c-peptide (>0,1 nmol/L)
Estimated glomerular filtration rate (GFR) (Cystatin C) | At day 75
  Cystatin C value
Portal vein thrombosis | The day after infusion
  Assessment by per protocol ultrasound
Bleeding | From infusion until 2 hours post start of infusion
  will be assessed by hemoglobin and thrombocyte monitoring (important while portal vein catheter is in place and withdrawn (within first week).

OTHER OUTCOMES:
The percentage of loss of radioactivity in the liver field. | Within the first two hours after start of islet infusion.
  When logistically feasible. Determined by positron emission tomography (PET)-scan of 2-deoxy-27fluoro-D-glucose ((18F) (FDG)-labelled islets infused in the portal vein as assessed during treatment (only possible at the Uppsala site).
Effect of eculizumab on IBMIR | Post infusion
  Determined by coagulation activation (TAT)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tufveson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Dept of Surgical Sciences, Section of Transplantation Surgery, University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207
- [Background] Eich T, Eriksson O, Lundgren T; Nordic Network for Clinical Islet Transplantation. Visualization of early engraftment in clinical islet transplantation by positron-emission tomography. N Engl J Med. 2007 Jun 28;356(26):2754-5. doi: 10.1056/NEJMc070201. No abstract available. PMID 17596618
- [Background] Eich T, Eriksson O, Sundin A, Estrada S, Brandhorst D, Brandhorst H, Langstrom B, Nilsson B, Korsgren O, Lundgren T. Positron emission tomography: a real-time tool to quantify early islet engraftment in a preclinical large animal model. Transplantation. 2007 Oct 15;84(7):893-8. doi: 10.1097/01.tp.0000284730.86567.9f. PMID 17984843
- [Background] Moberg L, Johansson H, Lukinius A, Berne C, Foss A, Kallen R, Ostraat O, Salmela K, Tibell A, Tufveson G, Elgue G, Nilsson Ekdahl K, Korsgren O, Nilsson B. Production of tissue factor by pancreatic islet cells as a trigger of detrimental thrombotic reactions in clinical islet transplantation. Lancet. 2002 Dec 21-28;360(9350):2039-45. doi: 10.1016/s0140-6736(02)12020-4. PMID 12504401
- [Background] Bennet W, Sundberg B, Groth CG, Brendel MD, Brandhorst D, Brandhorst H, Bretzel RG, Elgue G, Larsson R, Nilsson B, Korsgren O. Incompatibility between human blood and isolated islets of Langerhans: a finding with implications for clinical intraportal islet transplantation? Diabetes. 1999 Oct;48(10):1907-14. doi: 10.2337/diabetes.48.10.1907. PMID 10512353
- [Background] Koh A, Senior P, Salam A, Kin T, Imes S, Dinyari P, Malcolm A, Toso C, Nilsson B, Korsgren O, Shapiro AM. Insulin-heparin infusions peritransplant substantially improve single-donor clinical islet transplant success. Transplantation. 2010 Feb 27;89(4):465-71. doi: 10.1097/TP.0b013e3181c478fd. PMID 20177350
- [Background] Eriksson O, Eich T, Sundin A, Tibell A, Tufveson G, Andersson H, Felldin M, Foss A, Kyllonen L, Langstrom B, Nilsson B, Korsgren O, Lundgren T. Positron emission tomography in clinical islet transplantation. Am J Transplant. 2009 Dec;9(12):2816-24. doi: 10.1111/j.1600-6143.2009.02844.x. Epub 2009 Oct 21. PMID 19845588
- [Background] Friberg AS, Brandhorst H, Buchwald P, Goto M, Ricordi C, Brandhorst D, Korsgren O. Quantification of the islet product: presentation of a standardized current good manufacturing practices compliant system with minimal variability. Transplantation. 2011 Mar 27;91(6):677-83. doi: 10.1097/TP.0b013e31820ae48e. PMID 21248660